CLINICAL TRIAL: NCT06370988
Title: Theta-Burst Stimulation for Bipolar Depression
Acronym: TRIBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4343
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Depression; Bipolar Disorder; Treatment- Resistant Bipolar Disorder; Type 2 Bipolar Disorder
Keywords: Transcranial Magnetic Stimulation; Repetitive Transcranial Magnetic Stimulation; rTMS; iTBS
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: This trial will use a multi-centre randomized controlled trial for individuals with treatment-resistant Bipolar Depression comparing iTBS applied to the left DLPFC with sham treatment and examining differences in efficacy and safety outcomes between groups over 6 weeks of treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: rTMS treatment will be delivered using the MagPro X100/R30 stimulator and use the Cool-B70 A/P coil (MagVenture, Farum, Denmark), a figure 8 coil with active cooling, in which both the sham and active coils are contained internally. Its symmetric design ensures there is no indication of which side is active or sham with only the side of the coil delivering the treatment differing. The sham coil has been designed in such a way that it produces a similar auditory experience as the active coil. To account for the tactile sensation of active stimulation, both treatment allocations will have scalp electrodes placed that deliver a weak electrical stimulation to mask this tactile sensation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham iTBS Stimulation (Sham Comparator): Administered once daily over 30 days, using a sham coil that reproduces auditory and tactile sensations of stimulation and has an identical external appearance. Each session will deliver 600 pulses of sham iTBS in triplet 50Hz bursts, repeated at 5Hz 2s on 8s off for a total time of ~3 minutes, 9 seconds at a target intensity of 120% of the subject's resting motor threshold.
  Interventions: Device: Sham iTBS Stimulation
- Active iTBS Stimulation (Experimental): Administered once daily over 30 days. Each session will deliver 600 pulses of active iTBS in triplet 50Hz bursts, repeated at 5Hz 2s on 8s off for a total time of ~3 minutes, 9 seconds at a target intensity of 120% of the subject's resting motor threshold.
  Interventions: Device: iTBS Stimulation

INTERVENTIONS:
Device: iTBS Stimulation — Fluid-Cooled B70 A/P Coil with either Magventure X100 or R30
  Arms: Active iTBS Stimulation
Device: Sham iTBS Stimulation — Fluid-Cooled B70 A/P Coil with either Magventure X100 or R30
  Arms: Sham iTBS Stimulation

SUMMARY:
The purpose of this trial is to determine if intermittent theta-burst stimulation (iTBS) can reduce the symptoms of depression in treatment-resistant bipolar disorder. To do this, some of the participants in this study will receive treatment with active iTBS stimulation, while others will receive sham iTBS stimulation. Participants will come for 30 days of either active iTBS or sham iTBS, with a 6-week follow-up period. Symptoms of depression (for determining treatment efficacy) and mania (for determining treatment safety) will be assessed using the 17-item Hamilton Rating Scale for Depression (HRSD-17) and the Young Mania Rating Scale (YMRS) every five treatments during the treatment course, and at 1 week and 6 week after treatment completion.

ELIGIBILITY:
Inclusion Criteria

The participant must meet all of the inclusion criteria to eligible for this clinical trial:

1. Must be deemed to have capacity to provide informed consent;
2. Must be an outpatient
3. Have a DSM 5 diagnosis of bipolar disorder (type I or II), current episode depressed confirmed by Mini-International Neuropsychiatric Interview version 7.0.2 (MINI);
4. Age 18-65;
5. failure to achieve a clinical response to ≥1 adequate treatment trial for bipolar depression based on the Antidepressant Treatment History Form - Short Form (ATHF-SF) OR unable to tolerate at least 2 separate inadequate treatment trials for bipolar depression;43
6. moderately severe depression with a score ≥ 15 on the PHQ-9;44
7. not currently experiencing a mixed or manic episode (YMRS ≤10);
8. no increase or initiation of psychotropic medication with intention of treating depressive symptoms in the 4 weeks prior to screening. This excludes targeted treatment of insomnia with trazodone, melatonin, low-dose doxepin [3-6mg], low-dose benzodiazepines [≤2mg lorazepam daily equivalent], non-benzodiazepine benzodiazepine receptor agonists, or orexin antagonists;
9. able to adhere to the treatment schedule;
10. pass the TMS adult safety screening questionnaire.45

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this clinical trial:

1. have a history of MINI diagnosis of a substance use disorder (other than nicotine and/or caffeine) within the last 3 months;
2. have a concomitant major unstable medical illness;
3. have active suicidal intent (assessed during HRSD-17 Item 3 and SSRS as imminent intent to act on specific plan, confirmed by psychiatric staff);
4. are pregnant or intend to get pregnant during the study;
5. have a lifetime MINI diagnosis of schizophrenia or schizoaffective disorder;
6. have psychotic symptoms within the current episode;
7. have a MINI anxiety disorder, trauma-related disorder, obsessive compulsive disorder, or personality disorder assessed by a study investigator to be primary and/or causing greater impairment than BD-DE;
8. failure of an adequate acute course of ECT as defined by ATHF-SF during the current episode;
9. have received any rTMS before due to potential to compromise blinding of treatment allocation;
10. have any clinically significant neurological disorder (e.g., recent major cerebrovascular accident), or any history of seizure except those therapeutically induced by ECT or with clear precipitant (e.g., febrile seizure of childhood, alcohol withdrawal, etc.);
11. have any intracranial implant (e.g., aneurysm clips, shunts, stimulators,) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
12. are participating in psychotherapy for less than 3 months. Patients will be permitted if they have been in stable treatment for at least 3 months prior to study entry, with no anticipated change in the frequency of therapeutic sessions, or focus of therapeutic sessions over the duration of the study;
13. are currently taking lorazepam >2 mg daily (or equivalent) due to the potential to limit rTMS efficacy;
14. are currently taking any dose of an anticonvulsant due to the potential to limit rTMS efficacy. If anticonvulsants have been discontinued prior to screening, at least 5 half-lives have elapsed until screening to allow sufficient drug clearance;
15. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Change on the 17-item Hamilton Rating Scale for Depression (HRSD-17) | From enrollment to 6 weeks post-treatment
  Change on the 17-item Hamilton Rating Scale for Depression (HRSD-17), ITT, 6 weeks (completion of treatment phase (30 txs)). The main effect of interest is the interaction term between time since starting treatment and treatment allocation. This analytic approach incorporates longitudinal depressive symptom assessments throughout the trial rather solely at treatment completion.

SECONDARY OUTCOMES:
Symptoms of Mania | From enrollment to 6 weeks post-treatment
  Safety of rTMS in BD-DE with respect to symptoms of mania, Young Mania Rating Scale (YMRS), Safety Outcomes, 6 weeks (completion of treatment phase (30 txs)). The main effect of interest is the interaction term between time since starting treatment and treatment allocation. This analytic approach incorporates longitudinal depressive symptom assessments throughout the trial rather solely at treatment completion.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No